CLINICAL TRIAL: NCT05971134
Title: The Effect of Acupressure Applied to Different Fistula Area on Fistula Needle Insert Pain: A Randomized Clinical Trial
Brief Title: Acupressure and Fistula Needle Insert Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Gülay Turgay, assistant professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Acupressure
Record Dates: First submitted 2023-07-18; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Disease Stage 5 (Disorder)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Intervention group 1 consisted of patients with brescia-cimino fistula Intervention group 2 consisted of patients with snuff-box fistula Intervention group 3 consisted of patients with antecubital fistula.
  Interventions: Behavioral: Acupreesure applied
- Control Group (No Intervention): Control group 1 consisted of patients with brescia-cimino fistula Control group 2 consisted of patients with snuff-box fistula Control group 3 consisted of patients with antecubital fistula.

INTERVENTIONS:
Behavioral: Acupreesure applied — Acupressure was applied to the LI4 acupuncture point for 3 minutes by the researcher for the intervention group
  Arms: experimental group

SUMMARY:
Introduction: This study was conducted to determine the effectiveness of acupressure application on Hegu (LI4) point on the severity of acute pain caused by fistula needle in patients with brescia-cimino, snuff-box and antecubital fistula.

Methods: This study was randomized control study which was conducted with 66 intervention and 65 control participants. The participants in the intervention group were divided into 3 groups according to the fistula area. Data were collected using Descriptive Information Form and pain scale.

DETAILED DESCRIPTION:
This study is determined that finger acupuncture at L14 point reduces the severity of pain felt by the patient during fistula needle insertion. Acute pain during puncture of arteriovenous fistula is a common problem in hemodialysis patients. Moreover, patients experience this acute pain three times a week. Accordingly, acupressure applied to the L4 acupuncture point can be considered as an effective, simple and low-cost non-pharmacological method to reduce acute pain during needle insertion in patients. Since this application is non-invasive and does not carry the risk of complications, it can be taught to patients and/or nurses to contribute to the management of acute pain. In addition, in this article, we examined the effect of acupressure applied only to the LI4 acupuncture point on pain intensity during fistula needle insertion, therefore, we suggest designing different studies with different acupuncture points (effective in reducing pain).

ELIGIBILITY:
Inclusion Criteria

18 years or older have brescia-cimino, snuff-box or antecubital fistula speak Turkish have hemodialysis(HD) treatment three times a week have not used analgesics in the last 6 hours had no pain who volunteered to participate in the study.

Exclusion Criteria With aneurysmatic fistula had soft tissue damage infection in extremities has coagulations and bleeding problems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale was used to determine the severity of acute pain experienced by patients during fistula needle insertion. | 1 week
  The pain severity of the patient is determined with the Numeric Rating Scale. NRS includes numbers from 0 to 10. The meaning of the number "0" on the scale is "I have no pain" and the number "10" means "I have very severity pain".

CONTACTS AND LOCATIONS:
Overall Officials: Assistant prof. GÜLAY TURGAY, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the article is published